CLINICAL TRIAL: NCT01008423
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Assess the Efficacy and Safety of Budesonide Foam (2 mg/25 mL BID for 2 Weeks, Followed by 2 mg/25 mL QD for 4 Weeks) Versus Placebo in Subjects With Active Mild to Moderate Ulcerative Proctitis or Proctosigmoiditis
Brief Title: Efficacy and Safety of Budesonide Foam for Participants With Active Mild to Moderate Ulcerative Proctitis or Proctosigmoiditis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BUCF3002
Record Dates: First submitted 2009-11-04; First posted 2009-11-05 (Estimated); Results first posted 2019-08-14 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-07

CONDITIONS: Proctitis; Proctosigmoiditis
Keywords: Proctitis; Proctosigmoiditis; Ulcerative; Salix; Budesonide foam; Budesonide; Rectal; Gastrointestinal; Colitis; UC; UP; UPS; Additional relevant MeSH terms:; Proctocolitis; Ulcer; Colitis, Ulcerative; Gastroenteritis; Gastrointestinal Diseases; Digestive System Diseases; Rectal Diseases; Intestinal Diseases; Colonic Diseases; Sigmoid Diseases; Pathologic Processes; Inflammatory Bowel Diseases; Bronchodilator Agents; Autonomic Agents; Peripheral Nervous System Agents; Physiological Effects of Drugs; Pharmacologic Actions; Anti-Asthmatic Agents; Respiratory System Agents; Therapeutic Uses; Glucocorticoids; Hormones; Hormones, Hormone Substitutes, and Hormone Antagonists; Anti-Inflammatory Agents
MeSH Terms: conditions — Proctitis; Proctocolitis; Ulcer; Colitis; Colitis, Ulcerative; Gastroenteritis; Gastrointestinal Diseases; Digestive System Diseases; Rectal Diseases; Intestinal Diseases; Colonic Diseases; Sigmoid Diseases; Pathologic Processes; Inflammatory Bowel Diseases | interventions — Budesonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Budesonide (Experimental): Participants who were diagnosed with active mild to moderate UP or UPS, will receive 2 milligrams (mg)/25 milliliter (mL) of budesonide foam, rectally twice daily for a period of 2 weeks followed by 2 mg/25 mL of budesonide foam, rectally once daily for a period of 4 weeks.
  Interventions: Drug: Budesonide
- Placebo (Placebo Comparator): Participants who were diagnosed with active mild to moderate UP or UPS will receive 25 mL of placebo matching to budesonide foam twice daily for a period of 2 weeks followed by once daily for a period of 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Budesonide — Budesonide will be administered as per the dose and schedule specified in the respective arm.
  Arms: Budesonide
Drug: Placebo — Placebo matching to budesonide will be administered as per the dose and schedule specified in the respective arm.
  Arms: Placebo

SUMMARY:
The purpose of this study is to establish the efficacy profile of rectally administered budesonide foam, as compared to an equivalent volume of rectally administered placebo foam over the same dosing schedule, in participants who present with a diagnosis of active, mild to moderate, ulcerative proctitis (UP) or ulcerative proctosigmoiditis (UPS). During the study, eligible participants will be allowed to maintain previously established oral 5-aminosalicylic acid (5-ASA) treatment at doses up to 4.8 grams/day (g/day).

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily sign written informed consent.
* Male or non-pregnant and non-lactating females.
* Confirmed diagnosis (by endoscopy procedure) of active, mild to moderate UP or UPS, with disease extending at least 5 centimeters (cm) but no further than 40 cm from the anal verge.
* Must possess a baseline MMDAI score between 5 and 10.

Exclusion Criteria:

* History or current diagnosis of Crohn's disease and indeterminate colitis.
* Prior gastrointestinal surgery except appendectomy and hernia.
* Concomitant active gastrointestinal disease or distortion of intestinal anatomy.
* History of diverticulitis, collagenous colitis, celiac disease, recurrent pancreatic or known gallbladder disease.
* Uncontrolled, previously diagnosed type 1 or 2 diabetes mellitus.
* Uncontrolled abnormal thyroid function.
* Unstable significant cardiovascular, endocrine, neurologic or pulmonary disease.
* Hemoglobin levels less than (<) 7.5 grams /deciliter (g/dL).
* History of sclerosing cholangitis, cirrhosis, or hepatic impairment.
* Renal disease manifested by greater than (>) 2.0 milligrams/deciliter (mg/dL) serum creatinine.
* History of avascular hip necrosis, active tuberculosis, ocular herpes simplex or ocular varicella zoster, malignant disease, and HIV or hepatitis B or C.
* Adrenal insufficiency.
* Active systemic or cutaneous infection or toxic megacolon, fistula, perforation or abscess.
* History of uncontrolled psychiatric disorders or seizure disorders.
* History of asthma requiring ongoing use of inhaled steroids.
* Recent history of drug or alcohol abuse.
* Positive stool test for bacterial pathogens, Clostridium difficile toxin, or ovum and parasites.
* Vaccination within 28 days prior to randomization.
* Allergies to budesonide or to any other items used in its preparation.
* Participation in another clinical trial in the past 30 days.
* Pregnant or at risk of pregnancy.
* Taking a prohibited medication. Some medications to treat UP/UPS are prohibited during participation in the study, including laxatives and anti-diarrhea medications; however, oral 5-ASA agents at doses up to 4.8 g/day and daily fiber supplements are allowed. Other medications (e.g., antibiotics, anti-seizure and anti-coagulant medicines) are also prohibited.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 2009-11-20 (Actual); Primary Completion 2013-03-18 (Actual); Study Completion 2013-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director — Bausch Health Companies
Locations (62):
- United States (62):
  - Dothan, Alabama
  - Mesa, Arizona
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Chula Vista, California
  - Garden Grove, California
  - Mission Hills, California
  - Monterey, California
  - Roseville, California
  - San Francisco, California
  - Lafayette, Colorado
  - Bristol, Connecticut
  - Hamden, Connecticut
  - Altamonte Springs, Florida
  - Cape Coral, Florida
  - Hialeah, Florida
  - North Miami Beach, Florida
  - Winter Park, Florida
  - Macon, Georgia
  - Marietta, Georgia
  - Suwanee, Georgia
  - Moline, Illinois
  - Davenport, Iowa
  - Topeka, Kansas
  - Metairie, Louisiana
  - Annapolis, Maryland
  - Hagerstown, Maryland
  - Prince Frederick, Maryland
  - Silver Springs, Maryland
  - Chesterfield, Michigan
  - Rochester, Michigan
  - Tupelo, Mississippi
  - St Louis, Missouri
  - Egg Harbor, New Jersey
  - Marlton, New Jersey
  - Great Neck, New York
  - Mineola, New York
  - New York, New York
  - North Massapequa, New York
  - Stony Brook, New York
  - Asheville, North Carolina
  - Fayetteville, North Carolina
  - Greensboro, North Carolina
  - Jacksonville, North Carolina
  - New Bern, North Carolina
  - Raleigh, North Carolina
  - Rocky Mount, North Carolina
  - Wilmington, North Carolina
  - Beachwood, Ohio
  - Tulsa, Oklahoma
  - Portland, Oregon
  - Germantown, Tennessee
  - Houston, Texas
  - La Porte, Texas
  - Pasadena, Texas
  - Plano, Texas
  - San Antonio, Texas
  - Ogden, Utah
  - West Valley City, Utah
  - Chesapeake, Virginia
  - Lynchburg, Virginia
  - Monroe, Wisconsin

REFERENCES:
- [Derived] Bosworth BP, Sandborn WJ, Rubin DT, Harper JR. Baseline Oral 5-ASA Use and Efficacy and Safety of Budesonide Foam in Patients with Ulcerative Proctitis and Ulcerative Proctosigmoiditis: Analysis of 2 Phase 3 Studies. Inflamm Bowel Dis. 2016 Aug;22(8):1881-6. doi: 10.1097/MIB.0000000000000860. PMID 27416045
- [Derived] Sandborn WJ, Bosworth B, Zakko S, Gordon GL, Clemmons DR, Golden PL, Rolleri RL, Yu J, Barrett AC, Bortey E, Paterson C, Forbes WP. Budesonide foam induces remission in patients with mild to moderate ulcerative proctitis and ulcerative proctosigmoiditis. Gastroenterology. 2015 Apr;148(4):740-750.e2. doi: 10.1053/j.gastro.2015.01.037. Epub 2015 Jan 30. PMID 25644096

RESULTS

PARTICIPANT FLOW:
Groups:
- Budesonide: Participants who were diagnosed with active mild to moderate ulcerative proctitis (UP) or ulcerative proctosigmoiditis (UPS), received 2 milligrams (mg)/25 milliliter (mL) of budesonide foam, rectally twice daily for a period of 2 weeks followed by 2 mg/25 mL of budesonide foam, rectally once daily for a period of 4 weeks.
- Placebo: Participants who were diagnosed with active mild to moderate UP or UPS received 25 mL of placebo matching to budesonide foam twice daily for a period of 2 weeks followed by once daily for a period of 4 weeks.
Period: Overall Study
Arm/Group | Budesonide | Placebo
Started | 134 | 147
Received at Least 1 Dose of Study Drug | 134 | 147
Completed | 115 | 125
Not Completed | 19 | 22
Not completed — Adverse Event | 13 | 6
Not completed — Withdrawal by Subject | 4 | 7
Not completed — Lost to Follow-up | 0 | 2
Not completed — Low Cortisol | 0 | 1
Not completed — Lack of Efficacy | 0 | 5
Not completed — Disease Extent 70 centimeters (cm) | 1 | 0
Not completed — Personal Conflict | 1 | 0
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants.
Groups:
- Budesonide: Participants who were diagnosed with active mild to moderate UP or UPS, received 2 mg/25 mL of budesonide foam, rectally twice daily for a period of 2 weeks followed by 2 mg/25 mL of budesonide foam, rectally once daily for a period of 4 weeks.
- Total: Total of all reporting groups
Arm/Group | Budesonide | Placebo | Total
Number analyzed (Participants) | 134 | 147 | 281
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.3 (13.47) | 41.9 (13.27) | 43.0 (13.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 84 | 156
  Male | 62 | 63 | 125
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 17 | 32
  Not Hispanic or Latino | 119 | 130 | 249
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 11 | 8 | 19
  White | 119 | 135 | 254
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Remission
Description: Remission was a combined assessment of clinical and endoscopic variables, defined as an endoscopy score of less than or equal to (<=) 1, a rectal bleeding score of 0, and an improvement or no change from baseline in stool frequency subscales of the Modified Mayo Disease Activity Index (MMDAI) at the end of 6 weeks of treatment. MMDAI was used to assess the overall disease activity for each participant. MMDAI evaluated 4 indices: stool frequency, rectal bleeding, physician's global assessment (PGA) and endoscopy findings each on a scale of 0 to 3 with a maximum total score of 12. Stool frequency MMDAI subscore ranged from 0-3, where 0 indicated normal number of stools per day and 3 indicated 5 or more stools than normal. Rectal bleeding MMDAI subscore ranged from 0-3, where 0 indicated no blood seen and 3 indicated blood alone passed. Endoscopy MMDAI subscore ranged from 0-3, where 0 indicated normal or inactive disease and 3 indicated severe disease (spontaneous bleeding, ulceration).
Time Frame: Week 6
Population: ITT population included all randomized participants. Missing data was imputed using last observation carried forward (LOCF) method.
Measure: Number; unit: percentage of participants
Arm/Group | Budesonide | Placebo
Number analyzed (Participants) | 134 | 147
percentage of participants | 44.0 | 22.4
Statistical Analysis 1: Comparison: Budesonide vs Placebo; The logistic regression test was used to test for a difference in the percentages between the 2 treatment arms after adjusting for analysis center (country); Test type: Superiority; p < 0.0001, Regression, Logistic — Threshold for significance at 0.05 level

2. Secondary Outcome: Percentage of Participants Who Achieved a Rectal Bleeding MMDAI Subscale Score of 0 at End of Week 6
Description: The MMDAI was used to assess the overall disease activity for each participant. The MMDAI evaluated 4 indices:stool frequency, rectal bleeding, physician's global assessment and endoscopy findings each on a scale of 0 to 3 with a maximum total score of 12. Rectal bleeding MMDAI subscore ranged from 0-3, where 0 indicated no blood seen and 3 indicated blood alone passed. Missing data was imputed using LOCF method.
Time Frame: Week 6
Population: ITT population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Budesonide | Placebo
Number analyzed (Participants) | 134 | 147
percentage of participants | 50.0 | 28.6

3. Secondary Outcome: Number of Scheduled Assessments With Rectal Bleeding Responder Classification
Description: The MMDAI was used to assess the overall disease activity for each participant. The MMDAI evaluated 4 indices: stool frequency, rectal bleeding, PGA and endoscopy findings each on a scale of 0 to 3 with a maximum total score of 12. Rectal bleeding MMDAI subscore ranged from 0-3, where 0 indicated no blood seen and 3 indicated blood alone passed. Percentage of participants who were rectal bleeding responder at scheduled assessments were reported. Rectal bleeding responders were defined as those participants who achieved a rectal bleeding MMDAI subscale score of 0 during the treatment period. Missing data was imputed using LOCF method.
Time Frame: Weeks 1, 2, 4, and 6
Population: ITT population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Budesonide | Placebo
Number analyzed (Participants) | 134 | 147
percentage of participants
  Responder at 1 assessment | 8.2 | 18.4
  Responder at 2 assessment | 16.4 | 17.0
  Responder at 3 assessment | 21.6 | 7.5
  Responder at 4 assessment | 13.4 | 2.0

4. Secondary Outcome: Percentage of Participants Who Achieved an Endoscopy MMDAI Subscale Score of 0 or 1 at End of Week 6
Description: The MMDAI was used to assess the overall disease activity for each participant. The MMDAI evaluated 4 indices: stool frequency, rectal bleeding, physician's global assessment and endoscopy findings each on a scale of 0 to 3 with a maximum total score of 12. Endoscopy subscale ranged from 0-3, where 0 = normal or inactive disease, 1 = mild disease, 2 = moderate disease and 3 = severe disease (spontaneous bleeding, ulceration). Percentage of participants with normal or mild disease have been presented in this outcome measure. Missing data was imputed using LOCF method.
Time Frame: Week 6
Population: ITT population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Budesonide | Placebo
Number analyzed (Participants) | 134 | 147
percentage of participants | 56.0 | 36.7

5. Secondary Outcome: Percentage of Participants Who Achieved a Score of 0 for Rectal Bleeding Subscale and a Combined Score of <=2 for Bowel Frequency (BF) and Physician's Global Assessment (PGA) in the MMDAI Subscales at End of Week 6
Description: The MMDAI was used to assess the overall disease activity for each participant. The MMDAI evaluated 4 indices: stool frequency, rectal bleeding, PGA and endoscopy findings each on a scale of 0 to 3 with a maximum total score of 12. Rectal bleeding subscore ranged from 0-3, where 0 indicated no blood seen and 3 indicated blood alone passed. BF subscore ranged from 0-3, where 0 indicated normal number of stools per day and 3 indicated 5 or more stools than normal. PGA subscore ranged from 0-3, where 0 indicated normal disease and 3 indicated severe disease. Missing data was imputed using LOCF method.
Time Frame: Week 6
Population: ITT population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Budesonide | Placebo
Number analyzed (Participants) | 134 | 147
percentage of participants | 46.3 | 23.8

6. Secondary Outcome: Percentage of Participants Who Achieved an MMDAI Total Score of <= 3 With Greater Than or Equal to (>=2) Points of Improvement From Baseline at the End of Week 6
Description: The MMDAI was used to assess the overall disease activity for each participant. The MMDAI evaluated 4 indices: stool frequency, rectal bleeding, PGA and endoscopy findings each on a scale of 0 to 3 with a maximum total score of 12. Rectal bleeding subscore ranged from 0-3, where 0 indicated no blood seen and 3 indicated blood alone passed. BF subscore ranged from 0-3, where 0 indicated normal number of stools per day and 3 indicated 5 or more stools than normal. PGA subscore ranged from 0-3, where 0 indicated normal and 3 indicated severe disease. Endoscopy subscore ranged from 0-3, where 0 indicated normal and 3 indicated severe disease. MMDAI total score ranged from 0-12, where higher score indicated severe disease. Missing data was imputed using LOCF method.
Time Frame: Week 6
Population: ITT population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Budesonide | Placebo
Number analyzed (Participants) | 134 | 147
percentage of participants | 49.3 | 28.6

7. Secondary Outcome: Percentage of Participants Who Achieved Improvement of >=1 Point From Baseline in the MMDAI Endoscopy Subscale Score at End of Week 6
Description: The MMDAI was used to assess the overall disease activity for each participant. The MMDAI evaluated 4 indices: stool frequency, rectal bleeding, PGA and endoscopy findings each on a scale of 0 to 3 with a maximum total score of 12. Endoscopy subscore ranged from 0-3, where 0 = normal or inactive disease, 1 = mild disease (erythema, decreased vascular pattern), 2 = moderate disease (marked erythema, absent vascular pattern, friability, erosions), and 3 = severe disease (spontaneous bleeding, ulceration). Missing data was imputed using LOCF method.
Time Frame: Week 6
Population: ITT population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Budesonide | Placebo
Number analyzed (Participants) | 134 | 147
percentage of participants | 57.5 | 38.8

8. Secondary Outcome: Percentage of Participants Who Achieved Improvement of >=1 Point From Baseline in the MMDAI Rectal Bleeding Subscale Score at End of Week 6
Description: The MMDAI was used to assess the overall disease activity for each participant. The MMDAI evaluated 4 indices: stool frequency, rectal bleeding, PGA and endoscopy findings each on a scale of 0 to 3 with a maximum total score of 12. Rectal bleeding MMDAI subscore ranged from 0-3, where 0 = no blood seen, 1 = streaks of blood with stool less than half the time, 2 = obvious blood with stool most of the time, and 3 indicated blood alone passed. Missing data was imputed using LOCF method.
Time Frame: Week 6
Population: ITT population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Budesonide | Placebo
Number analyzed (Participants) | 134 | 147
percentage of participants | 72.4 | 56.5

9. Secondary Outcome: Percentage of Participants Who Achieved >=3 Point Improvement From Baseline in the MMDAI Total Score Including Improvement of >=1 Point From Baseline in the MMDAI Rectal Bleeding Subscale Score and MMDAI Endoscopy Subscale at End of Week 6
Description: as for outcome 6
Time Frame: Week 6
Population: ITT population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Budesonide | Placebo
Number analyzed (Participants) | 134 | 147
percentage of participants | 53.7 | 34.0

10. Secondary Outcome: Mean Change From Baseline to Week 6 in MMDAI Total Score and Subscale Scores
Description: as for outcome 6
Time Frame: Baseline, Week 6
Population: ITT population included all randomized participants. Here, 'Number analyzed' signifies number of participants evaluable for specified categories.
Measure: Mean (Standard Deviation); unit: unit on a scale
Arm/Group | Budesonide | Placebo
Number analyzed (Participants) | 134 | 147
unit on a scale
  Bowel frequency score: Baseline | 1.7 (0.95) | 1.8 (0.89)
  Bowel frequency score: Change at Week 6: number analyzed (Participants) | 133 | 147
  Bowel frequency score: Change at Week 6 | -0.8 (0.99) | -0.5 (0.92)
  Rectal Bleeding score:Baseline | 2.1 (0.39) | 2.1 (0.38)
  Rectal Bleeding score: Change at Week 6: number analyzed (Participants) | 133 | 147
  Rectal Bleeding score: Change at Week 6 | -1.3 (0.97) | -0.9 (0.93)
  PGA score:Baseline | 2.0 (0.26) | 2.0 (0.31)
  PGA score: Change at Week 6: number analyzed (Participants) | 133 | 147
  PGA score: Change at Week 6 | -0.9 (0.91) | -0.6 (0.76)
  Endoscopy score:Baseline | 2.1 (0.33) | 2.1 (0.28)
  Endoscopy score: Change at Week 6 | -0.9 (0.92) | -0.5 (0.79)
  Total score:Baseline | 7.9 (1.25) | 8.0 (1.17)
  Total score: Change at Week 6: number analyzed (Participants) | 133 | 145
  Total score: Change at Week 6 | -3.8 (3.20) | -2.5 (2.72)

ADVERSE EVENTS:
Time Frame: From start of study drug up to Week 8
Description: Safety population included all randomized participants who were administered at least one dose of the study drug.
Arm/Group | Budesonide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/134 | 0/147
Serious Adverse Events (participants affected / at risk) | 3/134 | 0/147
Other Adverse Events (participants affected / at risk) | 57/134 | 54/147
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Budesonide (N=134) | Placebo (N=147)
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Acute generalised exanthematous pustulosis (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Budesonide (N=134) | Placebo (N=147)
Sinusitis (Infections and infestations) | 1 | 1
Pyrexia (General disorders) | 0 | 2
Lymph node abscess (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2
Urinary tract infection (Infections and infestations) | 3 | 3
Pain (General disorders) | 0 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Chills (General disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 3 | 2
Flatulence (Gastrointestinal disorders) | 0 | 3
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1
Proctitis ulcerative (Gastrointestinal disorders) | 0 | 2
Haemorrhoids (Gastrointestinal disorders) | 0 | 2
Colonic polyp (Gastrointestinal disorders) | 1 | 1
Colitis ulcerative (Gastrointestinal disorders) | 2 | 2
Acute sinusitis (Infections and infestations) | 0 | 1
Otitis media acute (Infections and infestations) | 0 | 1
Abdominal tenderness (Gastrointestinal disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Headache (Nervous system disorders) | 2 | 6
Nasopharyngitis (Infections and infestations) | 2 | 3
Gout (Metabolism and nutrition disorders) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 2
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 2
Aspartate aminotransferase increased (Investigations) | 2 | 3
Fatigue (General disorders) | 2 | 2
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0
Asthenia (General disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1
Bacteriuria (Infections and infestations) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 4
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 4
Leukocytosis (Blood and lymphatic system disorders) | 1 | 1
Blood bilirubin increased (Investigations) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Bacterial test positive (Investigations) | 1 | 2
Blood cortisol decreased (Investigations) | 21 | 6
Constipation (Gastrointestinal disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Weight increased (Investigations) | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Faecal incontinence (Gastrointestinal disorders) | 0 | 1
Urine ketone body present (Investigations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1
Chest discomfort (General disorders) | 1 | 1
Dysgeusia (Nervous system disorders) | 0 | 1
Macular hole (Eye disorders) | 0 | 1
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 1
Influenza like illness (General disorders) | 1 | 0
Gingival swelling (Gastrointestinal disorders) | 1 | 0
Micturition urgency (Renal and urinary disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0
Blood bicarbonate decreased (Investigations) | 1 | 0
Blood calcium decreased (Investigations) | 1 | 0
Blood glucose decreased (Investigations) | 1 | 0
Blood potassium decreased (Investigations) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Urine analysis abnormal (Investigations) | 1 | 0
White blood cells urine positive (Investigations) | 2 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 3 | 0
Respiratory tract infection viral (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0
White blood cell count increased (Investigations) | 1 | 0
Tension headache (Nervous system disorders) | 1 | 0
Burning sensation (Nervous system disorders) | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0
Alopecia effluvium (Skin and subcutaneous tissue disorders) | 1 | 0
Anal pruritus (Gastrointestinal disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Please contact Sponsor directly for additional information.